CLINICAL TRIAL: NCT01021839
Title: Bovine Carotid Artery Graft Revisited: A Prospective, Randomized Comparison of Bovine Carotid Artery and Expanded Polytetrafluoroethylene for Permanent Hemodialysis Access
Brief Title: Comparison of Bovine Carotid Artery and Expanded Polytetrafluoroethylene (ePTFE) for Permanent Hemodialysis Access
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Artegraft, Inc. (Industry)
Responsible Party: Tatsuo Kawai, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2006p-000081
Record Dates: First submitted 2009-11-18; First posted 2009-11-30 (Estimated); Last update posted 2009-11-30 (Estimated); Status verified 2009-11

CONDITIONS: Kidney Failure; Renal Dialysis
Keywords: renal dialysis; bioprosthesis; arteriovenous shunt; surgical
MeSH Terms: conditions — Renal Insufficiency; Arteriovenous Fistula

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bovine Carotid Artery Graft (Active Comparator)
  Interventions: Procedure: Grafts placement
- Expanded Polytetrafluoroethylene Grafts (Active Comparator)
  Interventions: Procedure: Grafts placement

INTERVENTIONS:
Procedure: Grafts placement — Graft placement (upper or lower extremity); surgical or radiographic revision as needed.
  Other Names: Artegraft

SUMMARY:
The investigators did a randomized control trial comparing bovine carotid artery grafts with ePTFE grafts for patients that need hemodialysis access. The goal of the study was to determine differences in primary and assisted patency rates and frequency of complications between these two types of grafts. The investigators' hypothesis was that bovine carotid artery grafts more closely mimic autologous tissue and therefore, would provide better patency and fewer complications.

DETAILED DESCRIPTION:
Objective: To understand how bovine carotid artery (BCA) grafts compare to cuffed polytetrafluoroethylene (ePTFE) grafts as conduits for hemodialysis access in terms of patency and complications.

Background: Many hemodialysis patients do not have adequate anatomy for native arteriovenous fistulas. In these patients, synthetic conduits remain the only option for permanent hemodialysis access. We sought to compare the standard cuffed ePTFE with bovine carotid artery grafts as this has not been undertaken since the 1970's.

Methods: Following Institutional Review Board approval, a prospective, randomized controlled trial was conducted enrolling 29 patients in the BCA group and 28 patients in the ePTFE group. Univariate and multivariate analysis was undertaken to understand factors that affect complications. Patency rates were calculated using the Kaplan-Meyer method.

ELIGIBILITY:
Inclusion Criteria:

* Chronic kidney disease stage 4 or 5, in need of hemodialysis access

Exclusion Criteria:

* Surgically suitable for a native arteriovenous fistula

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2006-04; Primary Completion 2009-02 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Primary and Assisted Patency | 6, 12, 18, 24 months

SECONDARY OUTCOMES:
patients were monitored for the following complications: thrombosis of the graft; graft infection; pseudoaneurysm formation; steal syndrome. | 6,12,18 and 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Tatsuo Kawai, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States